CLINICAL TRIAL: NCT01247493
Title: Multicenter, Phase 2 Clinical Trial Evaluating the Efficacy and Tolerability of Induction and Consolidation Chemotherapy Comprising Fludarabine, Cytarabine, and Attenuated-dose Idarubicin in Elderly Patients With AML(Acute Myeloid Leukemia)
Brief Title: Modified-FLAI Induction and Consolidation Chemotherapy in Elderly Patient With Acute Myeloid Leukemia (AML)
Acronym: m-FLAI
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Kim, Inho professor, SeoulNUH
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H-0704-029-205
Record Dates: First submitted 2010-11-17; First posted 2010-11-24 (Estimated); Last update posted 2010-11-24 (Estimated); Status verified 2010-11

CONDITIONS: Acute Myeloid Leukemia
Keywords: fludarabine; AML; Efficacy; tolerability
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — Induction Chemotherapy; fludarabine; Cytarabine; Idarubicin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: induction chemotherapy (fludarabine, cytarabine, idarubicin) — fludarabine, cytarabine, idarubicin

SUMMARY:
A phase II clinical trial evaluating the efficacy and tolerability of induction and consolidation chemotherapy comprising Fludarabine, cytarabine and attenuated-dose Idarubicin (modified-FLAI) in the elderly patients with acute myeloid leukemia.

ELIGIBILITY:
Inclusion Criteria:

* previously untreated AML (excluding acute promyelocytic leukemia)
* age greater than 60 years old
* ECOG PS (Eastern Cooperative Oncology Group Performance scale) less than 2
* adequate hepatic/ renal/ cardiac function

Exclusion Criteria:

* acute promyelocytic leukemia
* significant cardiac disease
* combined non-hematologic malignancy
* aleukemic leukemia (only granulocytic sarcoma)
* CNS (Central Nervous system) involvement
* significant comorbidity/ uncontrollable bleeding tendency

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Actual)
Dates: Start 2007-06; Primary Completion 2009-06 (Actual); Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
Complete remission rate
  Rate of complete remssion (CR) after two cycles of m-FLAI induction

SECONDARY OUTCOMES:
Rate of serious adverse events (SAE)
  Number of patients dying from SAE related to m-FLAI induction
Event Free Survival
  Event free survival defined as a period from study enrollment to death by from cause or relapse of disease after complete remission
overall survival
  Overall survival defined as a period from study enrollment to death from any cause
Predictive factors for Complete remission
  Compare complete remission rate according to existence of specific chromosome abnormality and Charlson comorbidity index to evaluate predicative impact of these factors.

CONTACTS AND LOCATIONS:
Overall Officials: Inho Kim, Principal Investigator — professor
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

REFERENCES:
- [Derived] Kim I, Koh Y, Yoon SS, Park S, Kim BK, Kim DY, Lee JH, Lee KH, Cheong JW, Lee HK, Kim SH, Kim H, Joo YD, Lee SM, Won JH, Park SK, Hong DS, Kim SH, Sohn SK, Kim CS, Park E, Kim MK, Park MR, Lee JH, Min YH; Korean Society of Hematology AML/MDS working party. Fludarabine, cytarabine, and attenuated-dose idarubicin (m-FLAI) combination therapy for elderly acute myeloid leukemia patients. Am J Hematol. 2013 Jan;88(1):10-5. doi: 10.1002/ajh.23337. Epub 2012 Oct 17. PMID 23077109